CLINICAL TRIAL: NCT05865574
Title: A Randomized, Double-blind, Single-dose, Parallel Two-arm Study to Compare the Pharmacokinetics and Safety of BAT1706 Injection From Different Manufacturing Batches (by New Process and Old Process) in Healthy Subjects
Brief Title: A Comparative Pharmacokinetic Study to Evaluate Different Manufacturing Batches of BAT1706 Injection
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BAT-1706-004-CR
Record Dates: First submitted 2023-04-28; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-03

CONDITIONS: Healthy Men

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAT1706（New Process） (Experimental): Drug: BAT1706
  1 mg/kg, the corresponding volume of bulk solution should be drawn according to the actual body weight of the subject, diluted to 100 mL with 0.9% sodium chloride solution, and administered by intravenous drip
  Interventions: Drug: BAT1706 Injection
- BAT1706（Old Process） (Active Comparator): Drug: BAT1706
  1 mg/kg, the corresponding volume of bulk solution should be drawn according to the actual body weight of the subject, diluted to 100 mL with 0.9% sodium chloride solution, and administered by intravenous drip
  Interventions: Drug: BAT1706 Injection

INTERVENTIONS:
Drug: BAT1706 Injection — 1 vial/carton, 400 mg/16 mL/vial
  Other Names: BAT1706

SUMMARY:
This is a randomized, double-blind, single-dose, parallel two-arm study to compare the pharmacokinetics, safety, and immunogenicity of BAT1706 Injection from different manufacturing batches (by new process and old process) in healthy male subjects.

DETAILED DESCRIPTION:
A total of 38 subjects are planned to be enrolled and randomized in a 1: 1 ratio to receive a single intravenous drip of BAT1706 Injection (by old process) or BAT1706 Injection (by new process) at 1 mg/kg body weight.

A 7-day screening period will be set up for this study. Subjects will be admitted to the hospital 1 day pre-dose (Day -1) and discharged after completing relevant observations and assessments 24 h post-dose. After discharge, subjects should return to the hospital for 12 follow-up visits according to the requirements of this study, on Days 3, 4, 5, 8, 11, 15, 22, 29, 36, 43, 57 and 71 post-dose.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged between 18 and 45 years with body mass index (BMI) between 18.0 and 28.0 kg/m2 and body weight between 50 and 100 kg (inclusive);
2. Subjects for whom the results of physical examination, vital signs, 12-lead ECG, and laboratory tests are normal or abnormal without clinical significance;
3. Subjects who do not smoke, or smoke no more than 5 cigarettes per day for < 10 years;
4. Subjects who agree to use effective contraception (including but not limited to: hormonal contraception, physical contraception, or abstinence) from the time of signing the informed consent form until 6 months after intravenous drip of the study drug;
5. Subjects who are willing and able to follow the visits, treatments, laboratory tests, and other relevant procedures specified in this study.

Exclusion Criteria:

1. Subjects who have previous or current clinically significant gastrointestinal disorder (including diverticulitis, gastric ulcer), renal disorder, liver disorder, cardiovascular disorder, hematological disorder, lung disorder, nervous system disorder, metabolic disorder (including known diabetes mellitus), psychosis, or allergic disease (excluding mild asymptomatic seasonal allergy) at screening/enrollment, and in the opinion of the investigator, are not suitable for participation in this clinical study;
2. Subjects who have psychiatric disorders, or in the opinion of the investigator, are not suitable for participation in this clinical study (e.g., he is considered unable to understand or follow the relevant requirements of the study, or some of his existing conditions may result in additional risks associated with participation in this study);
3. Subjects who have previous or current clinically significant allergies (excluding mild asymptomatic seasonal allergy); or subjects who have known or suspected allergy or hypersensitivity to any component of the study drug; or subjects who have known or suspected hypersensitivity to Chinese hamster ovary cell products or other recombinant human or humanized antibodies;
4. Subjects who have a tendency to haemorrhage or thrombosis, or have a history of non-traumatic haemorrhage with appropriate clinical treatment, or have a history of thrombosis, or have any disease that may increase the risk of haemorrhage or thrombosis (e.g., abnormal coagulation, thrombocytopenia, or INR > 1.5);
5. Subjects who have any previous malignancy including lymphoma, leukemia, and skin cancer;
6. Subjects who have abnormal and clinically significant ECG (as judged by the investigator), or corrected QT interval according to Bazett's formula > 470 ms (Bazett's formula: Q-Tc = QT/(R-R)0.5, where R-R represents the interval between two R waves in s);
7. Subjects who have a history of hypertension, or systolic blood pressure > 145 mmHg or diastolic blood pressure > 95 mmHg at screening/enrollment;
8. Subjects who have clinically significant chronic or acute infection at screening/enrollment; or have any positive result for HBV surface antigen, HCV antibody, HIV antibody, and treponema pallidum antibody at screening;
9. Subjects who have previously used Bevacizumab or VEGF-targeting agents;
10. Subjects who have used any biological product within 3 months prior to enrollment, or have used any monoclonal antibody within 9 months prior to enrollment;
11. Subjects who have used prescription or over-the-counter drugs within 14 days prior to enrollment, or less than 5 half-lives have passed from the last dose to the dosing day of this study, whichever is longer;
12. Subjects who have used any Chinese herbal medicine within 14 days prior to enrollment;
13. Subjects who have participated in other drug clinical trials within 3 months prior to enrollment, or propose to participate in other drug clinical trials during this study;
14. Subjects who have received live virus vaccine within 12 weeks prior to screening, or plan to receive live virus vaccine during the study;
15. Subjects who have undergone major injury, surgery, or fracture within 4 weeks prior to enrollment, or propose to undergo surgery during the study;
16. Subjects who have donated blood or have blood samples > 400 mL collected as subjects within 3 months prior to screening, or plan to donate blood during the study;
17. Subjects who have a history of alcohol dependence, or have a positive alcohol test result at screening/baseline;
18. Subjects who have consumed alcoholic beverages within 48 h prior to enrollment;
19. Subjects who have a history of drug abuse, or have a positive drug abuse test result at screening/baseline;
20. Subjects who cannot follow the restrictions on smoking, alcohol consumption and concomitant medications for this study during the study;
21. Subjects who cannot stop high-intensity physical activities from the dosing day of the study drug until 30 days post-dose.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2024-01 (Estimated)

PRIMARY OUTCOMES:
AUC0-inf | Day1, 2, 3, 4, 5, 8,15, 22, 29, 36, 43, 57, 71
  Area under the plasma concentration-time curve from zero to infinity, AUC0-∞ = AUC0-t + Ct/λz
AUC0-t | Day1, 2, 3, 4, 5, 8,15, 22, 29, 36, 43, 57, 71
  Area under the blood concentration-time curve from time 0 to the last time point at which the concentration can be measured
Cmax | Day1, 2, 3, 4, 5, 8,15, 22, 29, 36, 43, 57, 71
  Maximum blood concentration
Tmax | Day1, 2, 3, 4, 5, 8,15, 22, 29, 36, 43, 57, 71
  Observed time to peak concentration
t1/2 | Day1, 2, 3, 4, 5, 8,15, 22, 29, 36, 43, 57, 71
  Elimination half-life t1/2 = 0.693/λz

SECONDARY OUTCOMES:
Adverse events | Day1, 2, 3, 4, 5, 8,15, 22, 29, 36, 43, 57, 71
  AE and SAE
Immunogenicity | Day1, 2, 3, 4, 5, 8,15, 22, 29, 36, 43, 57, 71
  Anti-drug antibody (ADA) positivity, ADA titer and neutralizing antibody (NAb) positivity for ADA.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Hu, Ph.D, Principal Investigator — The Second Hospital of Anhui Medical University
Locations (1):
- The Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui, China